CLINICAL TRIAL: NCT07342452
Title: A Prospective Pilot Study Comparing Immediate Combination Versus Sequential Treatment Using Injectable Poly-L-lactic Acid and Synchronous Ultrasound Parallel Beam Technology
Brief Title: Randomized Trial of Combination Treatment With Sofwave and Sculptra
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Molly A. Wanner, MD, Dermatologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P003217
Record Dates: First submitted 2026-01-05; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Skin Aging
Keywords: Laxity, Skin, Arm, Sofwave, Sculptra
MeSH Terms: interventions — New-Fill

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Sofwave and Sculptra same day (Active Comparator)
  Interventions: Device: Sofwave; Drug: Sculptra
- Sofwave and Sculptra one month apart (Active Comparator)
  Interventions: Device: Sofwave; Drug: Sculptra

INTERVENTIONS:
Device: Sofwave — parallel beam ultrasound on arm
Drug: Sculptra — Sculptra injection into arm

SUMMARY:
Evaluation of treatment on the upper arm with Sculptra and Sofwave on the same day versus Sofwave followed by Sculptra 1 month later.

DETAILED DESCRIPTION:
This is a prospective, single site, split-body, intra-individual comparison pilot study. Each subject serves as their own control. 13 subjects will be recruited for a goal of treatment 10 subjects. One upper extremity (proximal medial arm) will be randomized to receive immediate combination therapy with both injectable poly-L-lactic acid (PLLA, Sculptra®) and synchronous ultrasound parallel beam technology (Sofwave™) administered over the same day. The contralateral arm will undergo sequential therapy, with PLLA administered at baseline and synchronous ultrasound parallel beam treatment one month later (Treatment Visit #2, Day 30).

The study employs a randomized, split-body design to minimize inter-patient variability, with blinded investigator assessment of efficacy outcomes through assessment of standardized digital photographs and video of snap test (skin turgor test). taken during the Final Visit (Day 120).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥ 40 years old
2. Able to provide informed consent
3. Baseline level of upper arm skin flaccidity and volume loss as defined as type III or greater on the Arm Visual Analog Scale (Arm VAS) for aging

Exclusion Criteria:

* Prior treatment to the arms with a biostimulatory agent, energy-based device, or skin-tightening device within the past year.
* History of dermabrasion or deep peels involving the upper arms within the past year.
* History of prior surgery involving the upper arms.
* History of prior fat reduction procedures within the upper arms.
* History of keloids, hypertrophic scarring, or connective tissue disorders.
* Active dermatologic condition involving the treatment site.
* Active systemic or local infection or wounds at treatment site.
* History of lymphatic drainage problems involving the upper arms.
* Excessive subcutaneous fat in the upper arms as judged per the investigator.
* Use of immunosuppressive or anticoagulant/antiplatelet medications.
* Uncontrolled medical conditions interfering with wound healing or impacting bleeding.
* Use of weight loss medications or supplements within the month before the baseline visit.
* BMI ≥ 30 kg/m².
* Non-stable weight (>5% change) during the month prior to enrollment.
* Uncontrolled or current hormonal imbalance, including thyroid, pituitary, or androgen-related disorders.
* History of malignancy during the past 5 years.
* Implanted devices, such as pacemaker or defibrillator.
* Active pregnancy, recent pregnancy within the past 3 months, planning to become pregnant during the study period, and/or breastfeeding.
* History of heavy smoking during the past 10 years.
* History of substance abuse, mental dysfunction, or other factors limiting ability to cooperate with study procedures.
* Known allergy to any topical anesthetics or PLLA.
* Presence of metal implants or metallic foreign bodies within the treatment area (upper arms).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
GAIS skin laxity | From treatment to 3 months after treatment
  5-graded scale: worse; no change; improved; much improved; or very much improved.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States